CLINICAL TRIAL: NCT05147142
Title: Low Intensity Focused Ultrasound: a New Paradigm for Depression and Anxiety
Acronym: LIFU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ocean State Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB-2020-053
Record Dates: First submitted 2021-11-09; First posted 2021-12-07 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-04

CONDITIONS: Depression
Keywords: Functional Neuroimaging; Acoustic Stimulation; Focused Ultrasound
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind administration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Target Site Low Intensity Focused Ultrasound (Experimental): Low Intensity focused ultrasound of the target region. These are at a fundamental frequency = 650kHz, PRF = 10Hz, pulse width = 5ms, duty cycle = 5%; ISPTA.3 of 720 mW/cm2. As in prior studies, each sonication includes 10 pulsations, each lasting 30s, followed by 30s pause intervals; two 10-minute administrations provided per LIFU session.
  Interventions: Device: Low Intensity Focused Ultrasound
- Control Site Low Intensity Focused Ultrasound (Active Comparator): Low Intensity focused ultrasound of the control region. These are at a fundamental frequency = 650kHz, PRF = 10Hz, pulse width = 5ms, duty cycle = 5%; ISPTA.3 of 720 mW/cm2. As in prior studies, each sonication includes 10 pulsations, each lasting 30s, followed by 30s pause intervals; two 10-minute administrations provided per LIFU session.
  Interventions: Device: Low Intensity Focused Ultrasound

INTERVENTIONS:
Device: Low Intensity Focused Ultrasound — Brainsonix BX Pulsar 1002
  Other Names: LIFU

SUMMARY:
Objective: Preliminary studies show that low intensity focused ultrasound (LIFU), a new type of non invasive brain stimulation, may be able to reach deep structures of the brain involved with depression and anxiety, that remain inaccessible using current forms of non-invasive brain stimulation with precision. In this study, the investigators will test if this technique can be used to change brain activity in areas that are connected to depression and anxiety symptoms. The primary objectives of this study are to test the safety and tolerability of LIFU, evaluate the feasibility of using LIFU to reduce brain activity, and evaluate the feasibility of simultaneous fMRI-LIFU. If the results of this study are positive, what the investigators learn will serve as a strong foundation for the future development of innovative treatments for a variety of psychiatric disorders.

Research Procedures: 25 veterans will be recruited. Visits will take place at the VA Providence Healthcare System. During some visits, healthy and patient participants may undergo clinical and research neuroimaging, neuropsychological testing, complete questionnaires, and participate in clinical/neurological assessments. Healthy veterans will not receive LIFU and will only attend 2 study visits. Patients are expected to attend up to 8 visits over 6 weeks. However, some may require up to 6 extended follow-ups after visits 5 or 8, in which case they would attend a total of 11 or 14 visits over 6 months. Two patient visits will include the LIFU application, following FDA safety guidelines. Patients will be assigned either to an experiment in which LIFU stimulation will be delivered immediately prior to a task or to an experiment in which stimulation will be delivered during the task. Within each experiment, patients will be assigned to first receive either LIFU stimulation to the study target or anatomical control. Study staff, but not participants will know which location is being targeted in case safety concerns arise. Safety assessments will be conducted at follow-up visits. A clinician will be available during LIFU administration /follow-up visits. Assuming no injury or other concerns are present, patients will then repeat this process again, receiving stimulation targeting other brain area not previously selected.

ELIGIBILITY:
US military Veterans

Inclusion Criteria:

* Patients must meet DSM-5 criteria for major depressive disorder with and without anxiety symptoms
* Patients must also be symptomatic (i.e. symptom severity above clinical thresholds using standard rating scales) and, if relevant, stable treatment(s) for >6 weeks.

Exclusion Criteria:

* history of seizure disorder or serious neurologic illness including dementia
* structural or neurologic abnormalities present or in close proximity to sonication site for patients (e.g., clinically significant calcification as might be observed in Fahr disease)
* history of brain surgery, iv) pacemaker or implanted central nervous system device
* greater than mild traumatic brain injury, or any head injury within sixty days of participation
* greater than moderate alcohol or substance use disorders (last six months; excluding nicotine/caffeine)
* active use or withdrawal from alcohol or substances (assessed via breathalyzer/urine testing as indicated)
* metal in the head
* impediment to vision, hearing and/or hand use likely to interfere with assessments
* pregnant or lactating (assessed via pregnancy test)
* unable to follow protocols
* acute suicidality, defined as "Yes" on item 4 of the Columbia Suicide Severity Rating Scale (C-SSRS), (i.e., active suicidal ideation with some intent to act on thoughts), or any endorsement of item 5 (active ideation with specific plan and intent) or any actual, interrupted, aborted attempt or preparatory behavior within the past month.
* symptom threshold considered in the "very severe" range using standard rating scales will be excluded.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of LIFU-related adverse events as assessed by clinical MRI | up to 6 months post LIFU
  MRI safety and monitoring will be determined through the review of clinical MRIs. The clinical MRI will be used to detect possible LIFU-induced injury including edema or other injury and microvascular damage. While the investigators believe hyperacute injury to be unlikely, scans at 24 hours and 1-week will be used to monitor for later evolving injury. If injury is detected on any participant at any stage of the study, the investigators will halt all study procedures.
Incidence of LIFU-related adverse events as assessed by neurological examinations | up to 6 months post LIFU
  Neurological exams will be used to detect any possible LIFU-induced neurological changes.
Incidence of LIFU-related adverse events as assessed by neuropsychological testing | up to 6 months post LIFU
  The investigators will evaluate safety using standardized neuropsychological tests at baseline, 24 hours, and 1-week post LIFU. The Repeatable Battery for the Assessment of Neurocognitive Status (RBANS) will be used to measure attention, language, visuospatial/construction, immediate, and delayed memory and to measure any possible LIFU-induced changes across these domains.
Perfusion Arterial Spin Labeling (ASL) fMRI Signal throughout Brain | change from baseline to following sonication
  Perfusion ASL fMRI data will be collected before and after sonication. Analyses will assess the statistical relationship between ASL signal throughout the brain pre and post sonication.
BOLD fMRI Signal | change from baseline to following sonication
  BOLD data will be collected before, during, and following LIFU sonication. Analyses will assess any changes in BOLD signal in the brain following sonication.
Resting state functional connectivity | change from baseline to following sonication
  Resting state data will be collecting before, during, and following LIFU sonication. Analyses will assess any functional connectivity changes in the brain following sonication.

CONTACTS AND LOCATIONS:
Overall Officials: Noah S Philip, MD, Principal Investigator — VA Providence Healthcare System
Locations (1):
- VA Providence Healthcare System, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
data may be available via the NIMH Data Archive

REFERENCES:
- [Background] Korb AS, Shellock FG, Cohen MS, Bystritsky A. Low-intensity focused ultrasound pulsation device used during magnetic resonance imaging: evaluation of magnetic resonance imaging-related heating at 3 Tesla/128 MHz. Neuromodulation. 2014 Apr;17(3):236-41; discussion 241. doi: 10.1111/ner.12075. Epub 2013 May 10. PMID 23663228
- [Background] Monti MM, Schnakers C, Korb AS, Bystritsky A, Vespa PM. Non-Invasive Ultrasonic Thalamic Stimulation in Disorders of Consciousness after Severe Brain Injury: A First-in-Man Report. Brain Stimul. 2016 Nov-Dec;9(6):940-941. doi: 10.1016/j.brs.2016.07.008. Epub 2016 Jul 22. No abstract available. PMID 27567470
- [Background] Pasquinelli C, Hanson LG, Siebner HR, Lee HJ, Thielscher A. Safety of transcranial focused ultrasound stimulation: A systematic review of the state of knowledge from both human and animal studies. Brain Stimul. 2019 Nov-Dec;12(6):1367-1380. doi: 10.1016/j.brs.2019.07.024. Epub 2019 Jul 31. PMID 31401074
- [Background] Badran BW, Caulfield KA, Stomberg-Firestein S, Summers PM, Dowdle LT, Savoca M, Li X, Austelle CW, Short EB, Borckardt JJ, Spivak N, Bystritsky A, George MS. Sonication of the anterior thalamus with MRI-Guided transcranial focused ultrasound (tFUS) alters pain thresholds in healthy adults: A double-blind, sham-controlled study. Brain Stimul. 2020 Nov-Dec;13(6):1805-1812. doi: 10.1016/j.brs.2020.10.007. Epub 2020 Oct 24. PMID 33127579
- [Background] Philip NS, Arulpragasam AR. Reaching for the unreachable: low intensity focused ultrasound for non-invasive deep brain stimulation. Neuropsychopharmacology. 2023 Jan;48(1):251-252. doi: 10.1038/s41386-022-01386-2. No abstract available. PMID 35869281
- [Background] Arulpragasam AR, van 't Wout-Frank M, Barredo J, Faucher CR, Greenberg BD, Philip NS. Low Intensity Focused Ultrasound for Non-invasive and Reversible Deep Brain Neuromodulation-A Paradigm Shift in Psychiatric Research. Front Psychiatry. 2022 Feb 24;13:825802. doi: 10.3389/fpsyt.2022.825802. eCollection 2022. PMID 35280168